CLINICAL TRIAL: NCT06218602
Title: Pilot Trial of Fecal Microbiota Transplantation for Lymphoma Patients Receiving Axicabtagene Ciloleucel Therapy.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0581; NCI-2024-00282 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-01-11; First posted 2024-01-23 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Fecal Microbiota Transplantation; Drug Therapy; Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Will receive FMT therapy (both as a colonoscopy / FMT procedure and as capsules taken by mouth) plus the scheduled chemotherapy and CAR-T cell therapy.
  Interventions: Drug: Fecal Microbiota Transplantation; Procedure: Chemotherapy; Procedure: CAR-T Therapy
- Arm B (Experimental): Will receive no FMT therapy and only receive their scheduled chemotherapy and CAR-T cell therapy.
  Interventions: Procedure: Chemotherapy; Procedure: CAR-T Therapy

INTERVENTIONS:
Drug: Fecal Microbiota Transplantation — Given by PO
  Arms: Arm A
Procedure: Chemotherapy — Given by Infusion
Procedure: CAR-T Therapy — Given by Infusion

SUMMARY:
To find out if adding treatment with fecal microbiota transplantation (FMT) is effective at treating gut-related side effects of antibiotic treatment in participants who are receiving standard therapy with anti-CD19 chimeric antigen receptor T-cell (CAR-T cell) therapy.

DETAILED DESCRIPTION:
Primary Objectives

1. To assess the toxicity of combination of FMT with anti-CD19 Axicabtagene ciloleucel therapy and compare it with standard of care Arm B with anti-CD19 CAR-T arm
2. To assess the response in participants treated with the combination of FMT and Axicabtagene ciloleucel CAR T-cell therapy at day 30 and compare it with standard of care Arm B with anti-CD19 CAR-T arm.

Secondary Objectives

1. To assess PFS and OS among participants with and without FMT.
2. To assess changes in gut microbiome of lymphoma participants after FMT.
3. To assess dynamic changes in serum and stool metabolites after FMT.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age on the day of signing informed consent.
2. Histologically/cytologically confirmed diagnosis of B-cell lymphomas.
3. Is being planned to received FDA approved standard of care anti-CD19 Axicabtagene Ciloleucel.
4. Participants must have received or is receiving high-risk broad-spectrum antibiotics for minimum of two days within 180 days of scheduled Axicabtagene ciloleucel infusion. High-risk broad-spectrum antibiotics include carbapenems (meropenem, imipenem, doripenem), anti-pseudomonal antibiotics (cefepime, piperacillin-tazobactam, ceftazidime) or anaerobic antibiotics including metronidazole, clindamycin, amoxicillin-sulbactam.
5. An Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2. Evaluation of ECOG is to be performed within 7 days prior to the date of signing study consent.
6. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
7. Absolute neutrophil counts should be greater than 1000/ul at the time of administration of fecal enema.
8. Adequate hepatic function defined by a total bilirubin level ≤ 1.5 ≤ x the upper limit of normal (ULN)[except if Gilberts syndrome and then total bilirubin ≤ 3x is allowed], an AST, level ≤ 2.5 x ULN, and an ALT level ≤ 2.5 x ULN. If liver metastases are present, then AST and ALT levels must be ≤ 4 x ULN
9. Adequate renal function defined by an estimated creatinine clearance >30 mL/min according to the Cockcroft-Gault formula or by a creatinine clearance measurement from a 24-hour urine collection.
10. Highly effective contraception for both male and female subjects if the risk of conception exists. Highly effective contraception must be used 30 days prior to first study-drug administration, for the duration of trial treatment, and for at least for 12 months after treatment for females and 4 months after treatment for males. Should a female patient (or male participant's sexual partner) become pregnant or should either the female patient (or male participant's partner) suspect she is pregnant while the participant's study-participation is ongoing, the treating physician should be informed immediately.

Exclusion Criteria:

1. If participant received major surgery within last 4 weeks, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
2. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.
3. Has a diagnosis of primary immunodeficiency (excluding IgA deficiency).
4. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the study subject's best interest to participate, in the opinion of the treating investigator.
5. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
6. Pregnant or nursing women
7. For women of childbearing age, a serum pregnancy test will be required within 72 hours prior to enrollment. If the serum test is positive, patient will not be allowed to enroll in the trial.
8. Participants with history of irritable bowel disease and inflammatory bowel disease will be excluded from clinical trial.
9. Participants with difficulties in oral administration or at risk of aspiration (e.g., neurological issues)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Neeraj Saini, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Prasad R, Rehman A, Rehman L, Darbaniyan F, Blumenberg V, Schubert ML, Mor U, Zamir E, Schmidt S, Hayase T, Chang CC, McDaniel L, Flores I, Strati P, Nair R, Chihara D, Fayad LE, Ahmed S, Iyer SP, Wang M, Jain P, Nastoupil LJ, Westin J, Arora R, Turner J, Khawaja F, Wu R, Dennison JB, Menges M, Hidalgo-Vargas M, Reid K, Davila ML, Dreger P, Korell F, Schmitt A, Tanner MR, Champlin RE, Flowers CR, Shpall EJ, Hanash S, Neelapu SS, Schmitt M, Subklewe M, Francois-Fahrmann J, Stein-Thoeringer CK, Elinav E, Jain MD, Hayase E, Jenq RR, Saini NY. Antibiotic-induced loss of gut microbiome metabolic output correlates with clinical responses to CAR T-cell therapy. Blood. 2025 Feb 20;145(8):823-839. doi: 10.1182/blood.2024025366. PMID 39441941
- See also: MD Anderson Cancer Center — http://www.mdanderson.org